CLINICAL TRIAL: NCT05515406
Title: A Phase I, Open-label, Dose Escalation Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of ONO-7018 in Patients With Relapsed or Refractory NHL or CLL
Brief Title: A Study to Investigate the Safety, Tolerability, PK, PD, and Efficacy of ONO-7018 in Patients With R/R NHL or CLL
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ONO-7018-01
Record Dates: First submitted 2022-08-18; First posted 2022-08-25 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-07

CONDITIONS: Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell
Keywords: ONO-7018, MALT1 inhibitor, Lymphoma, Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma; Leukemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation Phase (Part 1) (Experimental): Up to 4 dose levels will be evaluated. Eligible patients will be assigned to a dose level cohort according to a traditional 3+3 dose escalation design.
  Interventions: Drug: ONO-7018
- Dose Expansion Phase (Part 2) (Experimental): Eligible patients will be assigned to the recommended dose level(s) selected from Part 1.
  Interventions: Drug: ONO-7018

INTERVENTIONS:
Drug: ONO-7018 — ONO-7018 tablet(s) are administered orally
  Arms: Dose Escalation Phase (Part 1)
Drug: ONO-7018 — ONO-7018 tablet(s) are administered orally
  Arms: Dose Expansion Phase (Part 2)

SUMMARY:
This is a Phase 1, open-label, multicenter study. This will be the first-in-human clinical study for ONO-7018 and will be conducted in two phases: a Dose Escalation Phase (Part 1) and a Dose Expansion Phase (Part 2).

DETAILED DESCRIPTION:
ONO-7018 is a selective inhibitor of mucosa associated lymphoid tissue protein 1 (MALT1) and is expected to exhibit antitumor activity in NHL and CLL. The purpose of this study is to determine the MTD and to evaluate the safety, tolerability, PK, pharmacodynamics (biomarkers), and efficacy of ONO-7018 in patients with relapsed or refractory NHL or CLL.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥ 18 years
2. Written informed consent by the patient or the patient's legally authorized representative
3. Patient with histologically/cytologically confirmed diagnosis of NHL or CLL
4. Patient with relapsed or refractory disease who has no available therapeutic options known to provide clinical benefit
5. Patient who has measurable disease
6. All acute toxic effects of any prior antitumor therapy, including investigational therapy, resolved to Grade ≤ 1 before the start of study therapy
7. Eastern Cooperative Oncology Group Performance Status 0 to 2
8. Adequate bone marrow, renal and hepatic functions

Exclusion Criteria:

1. History of lymphoid malignancy other than those allowed per inclusion criteria
2. Patient with central nervous system involvement
3. Patient with systemic and active infection
4. Any serious or uncontrolled medical disorder that may increase the risk associated with study participation or study treatment, or interfere with the interpretation of study results
5. Prior treatment with a MALT1 inhibitor
6. Patient receiving any other investigational drug within 4 weeks prior to study entry
7. Patient is unable to swallow tablets
8. Patient is found to be otherwise ineligible for the study by the investigator or sub investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2023-02-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Estimate of Maximum Tolerated Dose (MTD) | Up to 3 weeks
  MTD will be estimated based on Dose limiting toxicity (DLT) observed during the first 3 weeks of treatment
Incidence, causality, and severity of Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs) | Through study completion, an average of 1 year
  Adverse events with the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 used as a guide for the grading of severity.

SECONDARY OUTCOMES:
Plasma Concentration of ONO-7018 | Up to 48 weeks
  Plasma concentration will be assessed to evaluate Pharmacokinetics
Antitumor Activity of ONO-7018 (Overall Response Rate [ORR]) | Through study completion, an average of 1 year
  Antitumor activity of ONO-7018 as measured by ORR will be assessed according to the response criteria for Lymphoma.Lymphoma.
Antitumor Activity of ONO-7018 (Duration of Response [DOR]) | Through study completion, an average of 1 year
  Antitumor activity of ONO-7018 as measured by DOR will be assessed according to the response criteria for Lymphoma.
Antitumor Activity of ONO-7018 (Progression Free Survival [PFS]) | Through study completion, an average of 1 year
  Antitumor activity of ONO-7018 as measured by PFS will be assessed according to the response criteria for Lymphoma.
Antitumor Activity of ONO-7018 (Overall Survival [OS]) | Through study completion, an average of 1 year
  Antitumor activity of ONO-7018 as measured by OS will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Project Leader, Study Director — Ono Pharma USA Inc
Locations (10):
- United States (10):
  - Jonsson Comprehensive Cancer Center, Santa Monica, California
  - AMR Kansas City, Kansas City, Missouri
  - Leo Jenkins Cancer Center/ECU School of Medicine, Greenville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Baylor Scott & White Research Institute, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Northwest Medical Specialities, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: No